CLINICAL TRIAL: NCT03606239
Title: A Phase II Open-Label Multi-center Trial of Isotoxic Hypofractionated Chemoradiotherapy for NSCLC
Brief Title: NSCLC Isotoxic Hypofractionated Chemoradiotherapy
Acronym: IHRC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Xue Xiaoying, Director of Radiotherapy, The Second Hospital of Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSCLS isotoxic HypoRCT
Record Dates: First submitted 2018-06-27; First posted 2018-07-30 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: isotoxic; hypofractionated radiotherapy; Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- isotoxic hypofractionated group (Experimental): Hypofractionated radiation:
  1. Split mode: 3Gy/f. 2,Individualized prescriptions for different patients:
  (1) Spinal cord: 0%>45 Gy, and ≤2 Gy each time Lung: V20≤30%, V5≤65%, MLD≤16Gy Esophagus: highest dose ≤ 69Gy 3. Maximum limit: If the limit of any "A" is not reached, the maximum radiation dose is 69 Gy. The lowest radiation dose: 45Gy.
  Chemotherapy:
  Platinum-containing two-drug regimen: docetaxel + lobaplatin: Docetaxel 60 mg/m2, d1; Lobaplatin 30 mg/m2, d1; repeated every 28 days. The first cycle of chemotherapy started on the first day of radiotherapy.
  The same chemotherapy regimen is used up to 4 cycles as consolidation after the completion of radiotherapy.
  Interventions: Radiation: isotoxic hypofractionated group

INTERVENTIONS:
Radiation: isotoxic hypofractionated group — the normal tissue limits are uniform, such as: V20% ≤ 30%, spinal cord 0> 45Gy, etc., and used hypofractionated radiotherapy technology so that each patient received the maximum individualized radiation dose as possible，and the same time use the Platinum-containing drugs: docetaxel + lobaplatin Docetaxel 60 mg/m2, d1; Lobaplatin 30 mg/m2, d1, repeated every 28 days. The first cycle of chemotherapy started on the first day of radiotherapy.Consolidate chemotherapy up to 4 cycles after radiotherapy, as above.

SUMMARY:
Radiotherapy plays an important role in non-small cell lung cancer (NSCLC), and concurrent chemoradiation is considered to be the standard treatment for locally advanced NSCLC. However, due to the patient's physical condition, comorbidities and other reasons, only about 1/3 of patients can receive concurrent chemoradiation. Radiotherapy alone or sequential chemoradiation has become the treatment protocol for most patients. Hypofractionated radiotherapy can be used in NSCLC because it can shorten the over treatment time and may potentially reduce the effect of accelerated repopulation and obtain higher biological effective dose（BED）. So far, the vast majority of radiotherapy prescriptions have given a uniform dose of 60 Gy. This unified prescription dosage approach is completely inconsistent with the concept of precision treatment. The Netherlands MAASTRO put forward the concept of in silico radiotherapy prescription, that is: the normal tissue limits are uniform, such as: V20% ≤ 30%, spinal cord V0> 45Gy, etc., and each patient receives a different dose of radiation therapy. This radiation prescription could reach the limits of the normal tissue of every patient; if no one tissue limits were reached, the highest dose was set up to 79.2 Gy (1.8 Gy, BID). MAASTRO applied this "iso-toxic" radiotherapy prescription and used accelerated hyperfractionation technology so that each patient received the maximum individualized radiation dose as possible. We will integrate this concept with hypofractionated radiotherapy in order to further improve efficacy.

DETAILED DESCRIPTION:
Radiotherapy plays an important role in non-small cell lung cancer (NSCLC), and concurrent chemoradiation is considered to be the standard treatment for locally advanced NSCLC. However, due to the patient's physical condition, comorbidities and other reasons, only about 1/3 of patients can receive concurrent chemoradiation. Radiotherapy alone or sequential chemoradiation has become the treatment protocol for most patients. Hypofractionated radiotherapy can be used in NSCLC because it can shorten the total treatment time and may potentially reduce the effect of accelerated repopulation and obtain higher BED. So far, the vast majority of radiotherapy prescriptions have given a uniform dose of radiotherapy to all patients, regardless of individual factors such as tumor size, location, and adjacent vital organs, which may cause two consequences: First, small-volume tumors may, not receive enough radiation dose, resulting in a decrease in local control rate. Second, for large volumes of tumors or tumors adjacent to vital organs, even the "so-called" standard dose (60 Gy) may cause serious damage to normal tissues. This unified prescription dosage approach is completely inconsistent with the concept of precision treatment. The Netherlands MAASTRO put forward the concept of in silico radiotherapy prescription, that is: the normal tissue limits are uniform, such as: V20% ≤ 30%, spinal cord V0> 45Gy, etc., and each patient receives a different dose of radiation therapy.This radiation prescription could reach the limits of the normal tissue of every patient; if no one tissue limits were reached, the highest dose was set up to 79.2 Gy (1.8 Gy, BID). MAASTRO applied this "iso-toxic" radiotherapy prescription and used accelerated hyperfractionation technology so that each patient received the maximum individualized radiation dose as possible.From the model study to the long-term survival results, a series of encouraging results were achieved. The use of an individualized radiotherapy prescription based on iso-toxicity for the treatment of NSCLC in large-segment radiotherapy is expected to achieve: 1. For patients with small tumor volumes and no adjacent to vital organs, a higher radiation dose is given under safe conditions. 2. For patients with larger volumes of tumors or adjacent to vital organs, give safer doses.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological or cytological diagnosis of non-small cell lung cancer patients, the clinical stage using the eighth edition of American Joint Committee on Cancer（AJCC）, including stage III without resectable or who when SBRT/SABR are not suitable;
2. Age ≥ 18 years，≤ 75 years;
3. The expected survival period is ≥ 3 months;
4. Karnofsky performance status （KPS） score ≥ 60;
5. Normal blood account , liver and kidney function;
6. Forced expiratory volume in 1 second of 0.75 L or greater.

Exclusion Criteria:

1. Serious medical problems require hospitalization, include (but not limited to ): history of pulmonary fibrosis, previous myocardial infarction within 6 months, heart failure grade II and above, uncontrolled heart failure, uncontrolled chronic obstructive pulmonary disease （COPD）, uncontrolled diabetes .et al;
2. Esophageal invasion (cT4);
3. Others are not suitable for receiving radiotherapy and chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
radiation induced esophagitis and radiation induced pneumonitis | 2 years
  Number of participants with treatment-related severe adverse events：Grade IV radiation esophagitis, Grade III radiation esophagitis which results in interruption of radiotherapy for 7 days or more, and Grade III or above radiation pneumonitis

SECONDARY OUTCOMES:
time to disease progression (TTP) | 5 years
  Record the time from the start of enrollment to the objective progression of the tumor
progression-free survival(PFS) | 5 years
  Record the time from the start of enrollment to the progression of disease or death
overall survival (OS) | 5 years
  Record the time from the start of enrollment to progression or primary tumors
local control（LC） | 5 years
  record the proportion of no increase in primary tumor

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Ying Xue, Professor, Study Chair — The Second Hospital of Hebei Medical University; Qiang Lin, Professor, Study Director — North China Petroleum Bureau General Hospital, Hebei Medical University; Chao-Xing Liu, Professor, Study Director — No.1 Hospital of Shijiazhuang City
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Yes
After the publication of this study, we could share the IPD. However, this sharing is limited to academic research.
  Person to be contacted: Study Chair: Professor Xiao Ying Xue. Contact information: zyy_lq@petrochina.com.cn
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the publication of this study, we could share the IPD
Access Criteria: However, this sharing is limited to academic research. Person to be contacted: Study Chair: Professor Xiao Ying Xue.

REFERENCES:
- [Derived] Liu YE, Xue XY, Zhang R, Chen XJ, Ding YX, Liu CX, Qin YL, Li WQ, Ren XC, Lin Q. Study protocol: a multicentre, prospective, phase II trial of isotoxic hypofractionated concurrent chemoradiotherapy for non-small cell lung cancer. BMJ Open. 2020 Oct 23;10(10):e036295. doi: 10.1136/bmjopen-2019-036295. PMID 33099491